CLINICAL TRIAL: NCT04110626
Title: Realistic Evaluation of Expériences Animées, a School-based Intervention in Nouvelle Aquitaine
Acronym: ERIEAS
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2018/75
Record Dates: First submitted 2019-09-26; First posted 2019-10-01 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Addiction
Keywords: Addiction; Primary prevention; School-based programme
MeSH Terms: conditions — Behavior, Addictive | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Expériences Animées Programme: The Expériences Animées programme involves supervised short movies and talks with secondary school and high school pupils about the use of psychoactive substances.
  Interventions: Other: Questionnaires; Other: Non-directive Interviews

INTERVENTIONS:
Other: Questionnaires — The questionnaires are completed at the 3 survey times (T0, T1 and T2) by all pupils involved. Collected data are quantitative
Other: Non-directive Interviews — The interviews are conducted with 80 pupils/year randomly selected (i.e. 2 per class and 8 per establishment/year). Collected data are qualitative

SUMMARY:
The study is a realistic evaluation of the Expériences Animées school-based programme. The aim is to precisely characterize i) the effects in terms of alcohol and cannabis consumption, the use of health professionals in case of problematic use of those two substances; ii) the context and underpinning mechanisms triggered by the program in terms of changes of alcohol and cannabis representations and life skills development. This evaluation could allow to produce the key functions of the programme: how the intervention works, in which conditions.

DETAILED DESCRIPTION:
* Alcohol consumption represents the second main modifiable risk factor for cancer and the second preventable mortality cause in France, after tobacco use. It is mainly during adolescence, which corresponds to a period of integration with peers and a period of detachment from parents, that alcohol use starts. In France, alcohol remains the substance that adolescents most experiment with. A 2014 report shows that nearly half (49.4%) of first-year secondary school pupils have already tried an alcoholic drink and about one in seven secondary school pupils' reports having been drunk. The impact of cannabis consumption is wide as it can affect the social environment, the brain and the psychology of the consumers. Adolescence is a period during which the brain undergoes profound remodelling in areas that are high in cannabinoid receptors and that mediate cognitive control and emotion regulation. Therefore, childhood and adolescence are important stages of life on which preventive efforts may be focused, also because events occurring in the earliest stages of human development (before birth and during childhood) are known to be related to further risk for cancer, other chronic diseases and adult conditions.
* Among addiction prevention programmes, those that focus on life skills have been mentioned in the literature as being effective. In this context, the French organization "Association Ressources et Initiatives Addictions" (ARIA) has developed Expériences Animées programme (animated experiences) based on the above features, with the aim to help adolescents to change their representations and strengthen their life skills. This is a grassroots innovation. It has to be evaluated.
* The Expériences Animées programme involves supervised short movies and talks with secondary and high school pupils about the use of psychoactive substances. The movies are made specifically for the programme. The sessions are facilitated by two professionals including at least a clinical psychologist. In a given secondary/high school, one session per term is delivered for each class (40 classes). Three to five films are shown at each session. Each film aims to work on 2 to 3 life skills allowing to build protective behaviors against addictions. This programme is implemented since 2015.
* The investigators will collect quantitative and qualitative data to appraise the outcomes (O), mechanisms (M) and contextual elements (C), including the interventional elements) in order to verify the initial theories (hypothesis of causal pathways) by i) Questionnaires to collect outcomes in terms of consumption and health care, and some mechanisms: 2/ Non-directive interviews to collect mechanisms and contextual factors 3/ Observations to collect contextual elements during the sessions. The investigators will design the survey instruments in line with the initial middle-range theories identified.

ELIGIBILITY:
Inclusion Criteria:

Pupils :

* Pupils from the 10 secondary and high schools selected in the department of Charente, in 2nd and 5th years in 2019/2020 academic year,
* Pupils not opposite to participate and holders of parental authority not opposite to the participation of the child (no later than the day of inclusion)

Others :

* Non-opposition to participate of 3 Education professionals per establishment in the 10 secondary and high schools selected in the department of Charente,
* Non-opposition to participate of 2 session leaders,
* Non-opposition to participate of 3 funders.

Exclusion Criteria:

- Participants under legal protection

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pupils from 10 secondary and hugh schools in the department of Charente (France)
Sampling Method: Non-Probability Sample
Enrollment: 1026 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Daily, alcohol consumption | 3 years
  Alcohol consumption per day at study entry, after 1 year and after 2 years
Weekly, alcohol consumption | 3 years
  Alcohol consumption per week at study entry, after 1 year and after 2 years
Monthly, alcohol consumption | 3 years
  Alcohol consumption per month at study entry, after 1 year and after 2 years
Number of episodes of heavy drinking | 3 years
  An episode of heavy drinking : at least 5 drinks per occasion at study entry, after 1 year and after 2 years
Number of drunkenness episodes | 3 years
  Number of episodes at study entry, after 1 year and after 2 years
Weekly, cannabis consumption | 3 years
  Number of cannabis consumption per week at study entry, after 1 year and after 2 years
Monthly, cannabis consumption | 3 years
  Number of cannabis consumption per month at study entry, after 1 year and after 2 years
Yearly, cannabis consumption | 3 years
  Number of cannabis consumption per year at study entry, after 1 year and after 2 years
Number of consultation of a healthcare professional to discuss about a problematic use of alcohol and/or cannabis | 3 years
  Number of times at study entry, after 1 year and after 2 years

CONTACTS AND LOCATIONS:
Overall Officials: François ALLA, MD PhD, Principal Investigator — CIC1401-EC, Inserm-CHU de Bordeaux
Locations (1):
- CIC1401-EC - CHU de Bordeaux Centre Inserm U1219, Bordeaux, France

REFERENCES:
- [Derived] Martin-Fernandez J, Affret A, Martel E, Gallard R, Merchadou L, Moinot L, Termote M, Dejarnac V, Alla F, Cambon L. Realist evaluation of a theory-based life skills programme aiming to prevent addictive behaviours in adolescents: the ERIEAS study protocol. BMJ Open. 2020 Jun 29;10(6):e034530. doi: 10.1136/bmjopen-2019-034530. PMID 32601111